CLINICAL TRIAL: NCT05857670
Title: Women With BRCA1/2 Mutation: Guilt Feelings and Impact on Procreation Decision
Brief Title: Psyco Quality of Life and Procreation BRCA1/2
Acronym: QoL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1702/22
Record Dates: First submitted 2023-03-27; First posted 2023-05-12 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Genetic Predisposition
MeSH Terms: conditions — Breast Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Genetic predisposition to breast cancer — Guilt feelings about procreating

SUMMARY:
Women with breast and/or ovarian cancer or with a family history carried these pathologies can makeo genetic counseling in order to investigate whether they are carriers of the BRCA1/2 genetic mutation. This mutation exposes them to develop breast cancer from 50 to 80% and from 27 to 65% of developing ovarian cancer. BRCA1/2 mutations are inherited as an autosomal dominant manner and therefore there is a 50% probability of transmitting the mutation to the progeny. For this reason, women who have BRCA 1/2 mutation may be less likely to want children than those who test negative. The decision to have children could worry both for the probability to transfer the genetic mutation or because the parenthood could be compromised by the illness and/or by premature death. In previous studies, the psychological condition of patients with BRCA 1/2 mutations, with or without children, was only partially investigated. For this reason the main goal of the study is to deeply investigate the specific psychological condition, with particular attention to the guilt feelings on the possibility to transfer the genetic mutation to the progeny. In this wai it could be useful to development a therapeutic strategies aimed at the best adaptation of the patients to the new health condition.

ELIGIBILITY:
Inclusion Criteria:

* Women with BRCA1/2 mutation affected or not by breast neoplasm
* Women with BRCA1/2 mutation affected or not by breast neoplasm and with at least a son/daughter
* Women with at list middle school diploma
* Women available to do interviews

Exclusion Criteria:

* Women with other oncological pathology
* Women with cognitive deficient and/or inability to comply to the requirements of the study

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women with BRCA1/2 mutation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of feeling guilting | 24 monts
  * ISGR-15s
  * Il PFQ-2
  * PHQ-9

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - "Regina Elena" National Cancer Institute, Rome
  - Università dell'Insubria, Varese

IPD SHARING:
Plan to Share IPD: Undecided